CLINICAL TRIAL: NCT02906007
Title: A Phase I/II, Open-Label, Single Arm Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Bedaquiline (BDQ) Given in Combination With an Individualized Rifampin-Resistant Tuberculosis (RR-TB) Therapy in Infants, Children, and Adolescents With RR-TB Disease, Living With or Without HIV
Brief Title: Evaluating the Pharmacokinetics, Safety, and Tolerability of Bedaquiline in Infants, Children, and Adolescents With Multidrug-Resistant Tuberculosis, Living With or Without HIV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1108; 11884 (Registry Identifier: DAIDES Study ID Registry Number); IMPAACT P1108 (Other: NIAID)
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Results first posted 2025-03-21 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-03

CONDITIONS: Tuberculosis; HIV
MeSH Terms: conditions — Tuberculosis | interventions — bedaquiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (>=6 to < 18 years) (Experimental): Participants ≥30 kg: 400 mg once per day through the intensive PK sampling visit, then 200 mg three times per week on Monday, Wednesday, and Friday through the Week 24 visit Participants ≥15 to <30 kg: 200 mg once per day through the intensive PK sampling visit, then 100 mg three times per week on Monday, Wednesday, and Friday through the Week 24
  Interventions: Drug: Bedaquiline
- Cohort 2 (>=2 to < 6 years) (Experimental): Participants >7 to <30 kg: 200 mg once per day through the intensive PK sampling visit, then 100 mg three times per week on Monday, Wednesday, and Friday through the Week 24 visit
  Interventions: Drug: Bedaquiline
- Cohort 3 (>=0 to < 2 years) (Experimental): Participants >7 to <30 kg: 200 mg once per day through the intensive PK sampling visit, then 100 mg three times per week on Monday, Wednesday, and Friday through the Week 24 visit Participants ≥ 3 to ≤ 7 kg: 100 mg once per day through the intensive PK sampling visit, then 50 mg three times per week on Monday, Wednesday, and Friday through the Week 24 visit
  Interventions: Drug: Bedaquiline

INTERVENTIONS:
Drug: Bedaquiline — Participants received bedaquiline (BDQ) once per day through intensive PK sampling visit, then 3 times per week on Monday, Wednesday and Friday through the week 24 visit.
  Other Names: BDQ

SUMMARY:
P1108 was a Phase I/II, open-label, single-arm, exposure-controlled dose finding study of BDQ in infants, children, and adolescents living with and without HIV, with clinically diagnosed or bacteriologically confirmed rifampin-resistant tuberculosis (RR-TB). The study was designed to evaluate the PK, safety, and tolerability of BDQ over 24 weeks.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the pharmacokinetics (PK), safety, and tolerability of bedaquiline (BDQ) in combination with an individualized RR-TB therapy in infants, children, and adolescents with RR-TB disease, living with or without HIV.

This study was conducted among infants, children, and adolescents less than 18 years of age treated for clinically diagnosed or bacteriologically confirmed intra-thoracic (pulmonary) RR-TB and/or selected forms of extrathoracic RR-TB. Participants were assigned to cohorts based on age. Cohort 1 included children six years of age or older but less than 18 years of age; Cohort 2 included children two years of age or older but less than six years of age; and Cohort 3 included children 0 months of age and older but less than two years of age. Cohort 1 was divided into two weight bands, one for participants weighing 15 kg or more but less than 30 kg and one for participants weighing 30 kg or more. Cohort 2 included participants weighing greater than 7 kg. Cohort 3 included participants weighing at least 3 kg.

Study visits occured at enrollment (Day 0) and at Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, 32, 40, 48, 60, 72, 60, 72, and 96. Participants who exited the study before implementation of protocol Version 2.0 also had a study visit at Week 120. Participants in each cohort took BDQ once a day for approximately two weeks. For the next 22 weeks, BDQ was taken three times a week. Dosing for Cohorts 2 and 3 was based on data from Cohort 1.

Study visits included physical examinations, blood and urine collection, an electrocardiogram (ECG), medical history reviews, and other assessments.

ELIGIBILITY:
Inclusion Criteria:

* Parent/legal guardian willing and able to provide written informed consent for study participation; in addition, when applicable per local Institutional Review Board (IRB)/Ethics Committee (EC) policies and procedures, potential participant is willing and able to provide written assent for study participation.
* Age at enrollment:

  * Cohort 1: 6 years of age or older but younger than 18 years of age
  * Cohort 2: 2 years of age or older but younger than 6 years of age
  * Cohort 3: 0 months of age or older but younger than 2 years of age
* Weight at enrollment:

  * Cohort 1: At least 15 kg
  * Cohort 2: Greater than 7 kg
  * Cohort 3: At least 3 kg
* HIV status determined by testing requirements in the protocol.
* Either bacteriologically confirmed intrathoracic (pulmonary) RR-TB and/or any of the following forms of extrathoracic TB:

  * Peripheral TB lymphadenitis
  * Pleural effusion or fibrotic pleural lesions
  * Stage 1 TBM or clinically stable Stage 2A TBM*
  * Osteoarticular TB, including spinal TB
  * Other non-disseminated forms of TB disease OR

Probable RR-TB (or clinically diagnosed RR-TB) with the inclusion of intrathoracic and/or extrathoracic TB as listed below:

* A presumptive diagnosis of RR-TB based on well-documented clinical symptoms or signs of TB with chest radiological changes (in the case of intrathoracic TB), and/or any of the following extrathoracic disease manifestations:
* Peripheral TB lymphadenitis
* Pleural effusion or fibrotic pleural lesions
* Stage 1 TBM or clinically stable Stage 2A TBM
* Osteoarticular TB, including spinal TB
* Other non-disseminated forms of TB disease

More information on this criterion can be found in the protocol.

- Participant is on an RR-TB regimen as per local standard of care for at least seven days and not more than 12 weeks prior to entry, and tolerating the regimen well at entry, as determined by the site investigator based on available medical records.

Note: Participants may have received up to seven doses of non-study BDQ during the seven days prior to study enrollment. The date and dose amount of non-study BDQ doses must be available in medical records.

* For potential participants living with HIV: At least 14 days prior to entry, initiated an acceptable ART regimen defined as zidovudine/lamivudine/abacavir; NVP and two NRTIs; LPV/r and two NRTIs; an integrase class drug including dolutegravir or raltegravir with two NRTIs; or another regimen approved in advance by the Core Team.
* At entry, the participant has the following laboratory test results according to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (refer to the protocol for guidance on severity grading):
* Absolute neutrophil count (normal or grade 1)
* Creatinine (normal or grade 1)
* Aspartate Amino Transferase (AST) (normal or grade 1)
* Alanine Amino Transferase (ALT) (normal or grade 1)
* Total bilirubin (normal or grade 1) Note: Laboratory tests may be repeated during the screening period, with the latest results used for eligibility determination.
* If male and engaging in sexual activity that could lead to pregnancy of the female partner: At entry, participant agrees to use a barrier method of contraception (i.e., male condom), until four weeks after discontinuation of BDQ.
* If female and of reproductive potential, defined as having reached menarche and not having undergone a documented sterilization procedure (hysterectomy, bilateral oophorectomy, or salpingotomy): Negative pregnancy test at screening within five days prior to entry.
* If female, of reproductive potential (defined in the protocol), and engaging in sexual activity that could lead to pregnancy: At entry, participant agrees to avoid pregnancy and to use at least two of the following contraception methods from entry through completion of study follow-up: condoms, diaphragm or cervical cap, intrauterine contraceptive device (IUCD), hormonal-based contraception.
* For Cohort 3 participants less than six months of age: Gestational age at birth greater than or equal to 37 weeks as determined by the site investigator based on parent/guardian report and/or available medical records.

Exclusion Criteria:

* Has any documented or suspected clinically significant medical condition or any other condition (excluding HIV and TB) that, in the opinion of the site investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives.
* Known or presumed severe extrapulmonary manifestations of TB, including Stages 2B and 3 TBM as determined by the site investigator based on participant/parent/guardian report and/or available medical records.
* Participant is breastfeeding a child based on participant/parent/guardian report and/or available medical records.
* A significant cardiac arrhythmia that requires medication or a history of heart disease (heart failure, coronary artery disease) that increases the risk for Torsade de Pointes as determined by the site investigator based on participant/parent/guardian report and available medical records.
* QTcF interval greater than 460 ms (i.e., ECG mean triplicate value greater than 460 ms) at screening. Note: The centralized ECG read should be used during screening for eligibility determination.
* Clinically relevant ECG changes including but not limited to pathological Q-waves (defined as greater than 40 ms or depth greater than 0.4-0.5 mV); evidence of ventricular pre-excitation; evidence of complete or incomplete left bundle branch block or right bundle branch block; evidence of second or third degree heart block; intraventricular conduction delay with QRS duration greater than 120 ms; age-related bradycardia as defined by sinus rate less than lower limit as indicated in the protocol based on available medical records and centralized read of ECGs during screening.
* Known personal or family history of long QT syndrome as determined by the site investigator based on participant/parent/guardian report and/or available medical records.
* Within eight weeks prior to entry, participation in other clinical studies with investigational agents or devices, unless approved in advance by the Core Team.
* Taking any prohibited medications specified in the protocol within three days prior to entry based on participant/parent/guardian report and/or available medical records.

Ages: 0 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anneke Hesseling, M.D., Ph.D., Study Chair — Desmond Tutu TB Centre, Stellenbosch University
Locations (4):
- Les Centres GHESKIO Clinical Research Site (GHESKIO-INLR) CRS, Port-au-Prince, Haiti
- South Africa (3):
  - Sizwe CRS, Johannesburg, Gauteng
  - PHRU Matlosana CRS, Klerksdorp, North West
  - Desmond Tutu TB Centre - Stellenbosch University (DTTC-SU) CRS, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017, will be used in this study — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: "Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010" — https://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first enrollment to the study was in September 2017 and enrollment was completed in August 2023 with a total of 54 participants who initiated study drug. There enrollments were from one site in Haiti - Les Centres Gheskio INLR CRS, and three sites from South Africa - Desmond Tutu TB Center - Stellenbosch University, Sizwe CRS, and PHRU Matlosana CRS.
Groups:
- Cohort 1 (≥ 6 to < 18 Years): Participants ≥30 kg:
  400 mg once per day through the intensive PK sampling visit, then 200 mg three times per week on Monday, Wednesday, and Friday through the Week 24 visit
  Participants ≥15 to <30 kg:
  200 mg once per day through the intensive PK sampling visit, then 100 mg three times per week on Monday, Wednesday, and Friday through the Week 24 visit
- Cohort 2 (≥ 2 to < 6 Years): Participants >7 to <30 kg:
  200 mg once per day through the intensive PK sampling visit, then 100 mg three times per week on Monday, Wednesday, and Friday through the Week 24 visit
- Cohort 3 (≥ 0 to < 2 Years): Participants >7 to <30 kg:
  200 mg once per day through the intensive PK sampling visit, then 100 mg three times per week on Monday, Wednesday, and Friday through the Week 24 visit
  Participants ≥ 3 to ≤ 7 kg:
  100 mg once per day through the intensive PK sampling visit, then 50 mg three times per week on Monday, Wednesday, and Friday through the Week 24 visit
Period: Overall Study
Arm/Group | Cohort 1 (≥ 6 to < 18 Years) | Cohort 2 (≥ 2 to < 6 Years) | Cohort 3 (≥ 0 to < 2 Years)
Started | 18 | 18 | 18
Completed (Through 24 weeks of study treatment) | 17 | 18 | 17
Not Completed | 1 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Died | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 (≥ 6 to < 18 Years): Bedaquiline: Participants ≥30 kg:
  400 mg once per day through the intensive PK sampling visit, then 200 mg three times per week on Monday, Wednesday, and Friday through the Week 24 visit
  Participants ≥ 15 to <30 kg:
  200 mg once per day through the intensive PK sampling visit, then 100 mg three times per week on Monday, Wednesday, and Friday through the Week 24 visit
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (≥ 6 to < 18 Years) | Cohort 2 (≥ 2 to < 6 Years) | Cohort 3 (≥ 0 to < 2 Years) | Total
Number analyzed (Participants) | 18 | 18 | 18 | 54
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 12.7 [7.0 to 13.8] | 3.4 [2.8 to 4.4] | 1.2 [0.7 to 1.8] | 3.4 [1.8 to 7.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 9 | 30
  Male | 6 | 9 | 9 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black African | 15 | 10 | 15 | 40
  Coloured | 3 | 7 | 3 | 13
  Mixed | 0 | 1 | 0 | 1
HIV-1 status [Count of Participants; unit: Participants]
  not living with HIV | 13 | 17 | 16 | 46
  living with HIV | 5 | 1 | 2 | 8
Weight [Median (Inter-Quartile Range); unit: kilogram (kg)] | 36 [20 to 41] | 13 [11 to 15] | 9 [7 to 10] | 13 [10 to 20]
Height [Median (Inter-Quartile Range); unit: centimeter (cm)] | 151 [117 to 159] | 95 [86 to 100] | 74 [68 to 79] | 95 [79 to 117]
TB disease spectrum [Count of Participants; unit: Participants]
  Pulmonary TB (PTB) | 15 | 17 | 17 | 49
  Extra Pulmonary TB (EPTB) | 1 | 0 | 0 | 1
  PTB and EPTB | 2 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events of ≥ Grade 3 Severity
Description: At entry and follow-up, all lab results, signs and symptoms, and diagnoses were recorded. The core team reviewed and confirmed the sites assessment of event relatedness to study drug. An adverse event (AE) is any unfavorable and unintended sign, symptom, or diagnosis that occurs in a study participant during the conduct of the study REGARDLESS of the attribution. Adverse events are graded on a scale from 1-5: 1=mild, 2=moderate, 3=severe, 4= potentially life-threatening, 5=death. AE grading was per Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table V2.1).
Time Frame: Measured from entry through Week 24
Population: All participants enrolled in the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (≥ 6 to < 18 Years) | Cohort 2 (≥ 2 to < 6 Years) | Cohort 3 (≥ 0 to < 2 Years)
Number analyzed (Participants) | 18 | 18 | 18
percentage of participants | 38.9 [17.3 to 64.3] | 11.1 [1.4 to 34.7] | 83.3 [58.6 to 96.4]

2. Primary Outcome: Percentage of Participants With Adverse Events of ≥ Grade 3 Assessed by the Core Team to be at Least Possibly Related to the Study Drug
Description: At entry and follow-up, all lab results, signs and symptoms, and diagnoses were recorded. The core team reviewed and confirmed the sites assessment of event relatedness to study drug. An adverse event (AE) is any unfavorable and unintended sign, symptom, or diagnosis that occurs in a study participant during the conduct of the study REGARDLESS of the attribution. Adverse events are graded on a scale from 1-5: 1=mild, 2=moderate, 3=severe, 4= potentially life-threatening, 5=death. AE grading was per Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table V2.1.
Time Frame: Measured from entry through Week 24
Population: All participants enrolled in the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (≥ 6 to < 18 Years) | Cohort 2 (≥ 2 to < 6 Years) | Cohort 3 (≥ 0 to < 2 Years)
Number analyzed (Participants) | 18 | 18 | 18
percentage of participants | 5.6 [0.1 to 27.3] | 0 [0 to 18.5] | 0 [0 to 18.5]

3. Primary Outcome: Percentage of Participants Who Were Terminated From Study Treatment Due to a Drug-related Adverse Event
Description: as for outcome 2
Time Frame: Measured from entry through Week 24
Population: All participants enrolled in the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (≥ 6 to < 18 Years) | Cohort 2 (≥ 2 to < 6 Years) | Cohort 3 (≥ 0 to < 2 Years)
Number analyzed (Participants) | 18 | 18 | 18
percentage of participants | 0 [0 to 18.5] | 0 [0 to 18.5] | 0 [0 to 18.5]

4. Primary Outcome: Percentage of Participants Who Died
Description: At entry and follow-up, all lab results, signs and symptoms, and diagnoses were recorded. The core team reviewed and confirmed the sites assessment of event relatedness to study drug. An adverse event (AE) is any unfavorable and unintended sign, symptom, or diagnosis that occurs in a study participant during the conduct of the study REGARDLESS of the attribution. Adverse events are graded on a scale from 1-5: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death. AE grading was per Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table V2.0.
Time Frame: Measured from entry through Week 24
Population: All participants enrolled in the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 1 (≥ 6 to < 18 Years): Bedaquiline: Participants ≥30 kg:
  400 mg once per day through the intensive PK sampling visit, then 200 mg three times per week on Monday, Wednesday, and Friday through the Week 24 visit
  Participants ≥15 to <30 kg:
  200 mg once per day through the intensive PK sampling visit, then 100 mg three times per week on Monday, Wednesday, and Friday through the Week 24 visit
Arm/Group | Cohort 1 (≥ 6 to < 18 Years) | Cohort 2 (≥ 2 to < 6 Years) | Cohort 3 (≥ 0 to < 2 Years)
Number analyzed (Participants) | 18 | 18 | 18
percentage of participants | 5.6 [0.1 to 27.3] | 0 [0 to 18.5] | 0 [0 to 18.5]

5. Primary Outcome: Percentage of Participants With Unstable Dysrhythmias Requiring Hospitalization and Treatment
Description: At entry and follow-up, any participant who experienced unstable dysrhythmias that required hospitalization and treatment were considered as an adverse event. The core team reviewed and confirmed the sites assessment of event relatedness to study drug.
Time Frame: Measured from entry through Week 24
Population: All participants enrolled in the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (≥ 6 to < 18 Years) | Cohort 2 (≥ 2 to < 6 Years) | Cohort 3 (≥ 0 to < 2 Years)
Number analyzed (Participants) | 18 | 18 | 18
percentage of participants | 0 [0 to 18.5] | 0 [0 to 18.5] | 0 [0 to 18.5]

6. Primary Outcome: Percentage of Participants With Absolute Corrected QT Interval by Fridericia (QTcF) ≥ 500 Msec
Description: Evaluation of the Electrocardiogram (ECG) QTcF was performed per protocol. ECGs conducted at these visits should be performed in triplicate (if possible). Consultation with the protocol cardiologist was available and encouraged for any abnormal or equivocal ECG findings and/or questions related to cardiac toxicities and assessment. Participants were included if they had QTcF ≥ 500 msec at any study visit from entry to Week 24.
Time Frame: All participants had ECG performed at Screening and Entry visits and through week 24.
Population: All participants enrolled in the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (≥ 6 to < 18 Years) | Cohort 2 (≥ 2 to < 6 Years) | Cohort 3 (≥ 0 to < 2 Years)
Number analyzed (Participants) | 18 | 18 | 18
percentage of participants | 5.6 [0.1 to 27.3] | 0 [0 to 18.5] | 0 [0 to 18.5]

7. Primary Outcome: Geometric Mean of Area Under the Concentration Versus Time Curve (AUC0-24h or AUC0-168h) Bedaquiline
Description: PK parameter determined from plasma concentration-time profiles, dosing information and participant covariates using the final population PK model
  The final population PK model was developed using a nonlinear mixed effects model (NNMEM, version 7.5).
  * Developed a population PK model as part of the final PK analysis
  * Data used in the population PK analysis included the intensive PK visit (Week 1 or Week 2), sparse PK samples from Weeks 4, 8, 12, 16, 20, 24, etc,as available at time of final analysis (when all participants have at least Week 24 PK samples)
  * Estimated individual AUC values at given time points for each participant using the developed model
Time Frame: Intensive PK Week 1 or 2, Week 8, and Week 24, (if intensive then pre dose, and post dose at 2, 4, 6, 8 hours) and if not intensive then predose only.
Population: * Participants that have completed the intensive PK sampling collection and have at least one sample with measurable BDQ and M2 concentrations
  * For intensive PK (week 1 or 2) metrics: Participants with PK sampling that is not after a BDQ daily dose will be excluded
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*mg/L
Arm/Group | Cohort 1 (≥ 6 to < 18 Years) | Cohort 2 (≥ 2 to < 6 Years) | Cohort 3 (≥ 0 to < 2 Years)
Number analyzed (Participants) | 18 | 18 | 18
hour*mg/L
  Intensive PK (week 1 or 2) (AUC0-24): number analyzed (Participants) | 15 | 18 | 15
  Intensive PK (week 1 or 2) (AUC0-24) | 32.6 (59.8) | 56.5 (32.7) | 60.3 (52.1)
  Week 8 (AUC0-168h) | 121 (51.3) | 179 (19.4) | 194 (58.3)
  Week 24 (AUC0-168h): number analyzed (Participants) | 17 | 18 | 17
  Week 24 (AUC0-168h) | 125 (50.8) | 180 (20.3) | 202 (51.8)

8. Secondary Outcome: Percentage of Participants With Adverse Events ≥ Grade 3 Severity
Description: as for outcome 1
Time Frame: Measured through Week 96 or 72 weeks post BDQ discontinuation
Reporting Status: Not Posted, anticipated posting 2026-08

9. Secondary Outcome: Percentage of Participants With Adverse Events ≥ Grade 3 Severity Assessed by the Core Team to be at Least Possibly Related to the Study Drug.
Description: as for outcome 1
Time Frame: Measured through Week 96 or 72 weeks post BDQ discontinuation
Reporting Status: Not Posted, anticipated posting 2026-08

10. Secondary Outcome: Percentage of Participants With Absolute Corrected QT Interval by Fridericia (QTcF) ≥ 500 Msec
Description: as for outcome 6
Time Frame: Measured through Week 96 or 72 weeks post BDQ discontinuation
Reporting Status: Not Posted, anticipated posting 2026-08

11. Secondary Outcome: Percentage of Participants With Unstable Dysrhythmias Requiring Hospitalization and Treatment
Description: as for outcome 1
Time Frame: Measured through Week 96 or 72 weeks post BDQ discontinuation
Reporting Status: Not Posted, anticipated posting 2026-08

12. Secondary Outcome: Percentage of Participants Who Died
Description: as for outcome 1
Time Frame: Measured through Week 96 or 72 weeks post BDQ discontinuation
Reporting Status: Not Posted, anticipated posting 2026-08

13. Secondary Outcome: Geometric Mean of Area Under the Concentration Versus Time Curve (AUC0-24h or AUC0-168h) Bedaquiline Mono-desmethyl Metabolite (M2)
Description: as for outcome 7
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*mg/L
Arm/Group | Cohort 1 (≥ 6 to < 18 Years) | Cohort 2 (≥ 2 to < 6 Years) | Cohort 3 (≥ 0 to < 2 Years)
Number analyzed (Participants) | 18 | 18 | 18
hour*mg/L
  Intensive PK (Week 1 or 2) (AUC0-24): number analyzed (Participants) | 15 | 18 | 15
  Intensive PK (Week 1 or 2) (AUC0-24) | 9.14 (30.6) | 11.3 (50.2) | 8.63 (57.9)
  Week 8 (AUC0-168h) | 28.4 (40.1) | 41.4 (32.0) | 33.0 (56.6)
  Week 24 (AUC0-168h): number analyzed (Participants) | 17 | 18 | 17
  Week 24 (AUC0-168h) | 32.6 (39.6) | 45.0 (29.5) | 39.3 (48.3)

14. Secondary Outcome: Geometric Mean of Maximal Concentration (Cmax) Bedaquiline
Description: as for outcome 7
Time Frame: Intensive PK Week 1 or 2, Week 8, and Week 24, (if intensive then pre dose, and post dose at 2, 4, 6, 8 hours) and if not intensive then pre dose only.
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Cohort 1 (≥ 6 to < 18 Years) | Cohort 2 (≥ 2 to < 6 Years) | Cohort 3 (≥ 0 to < 2 Years)
Number analyzed (Participants) | 18 | 18 | 18
mg/L
  Intensive PK (Week 1 ir 2) (Cmax): number analyzed (Participants) | 15 | 18 | 15
  Intensive PK (Week 1 ir 2) (Cmax) | 2.16 (54.2) | 3.72 (34.8) | 4.22 (43.4)
  Week 8 (Cmax) | 1.92 (34.3) | 2.37 (20.5) | 2.73 (31.1)
  Week 24 (Cmax): number analyzed (Participants) | 17 | 18 | 17
  Week 24 (Cmax) | 2.01 (35.3) | 2.42 (19.3) | 2.66 (33.6)

15. Secondary Outcome: Geometric Mean of Maximal Concentration (Cmax) Bedaquiline Mono-desmethyl Metabolite (M2)
Description: PK parameter determined from plasma concentration-time profiles, dosing information and participant covariates using the final population PK model
Time Frame: as for outcome 14
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Cohort 1 (≥ 6 to < 18 Years) | Cohort 2 (≥ 2 to < 6 Years) | Cohort 3 (≥ 0 to < 2 Years)
Number analyzed (Participants) | 18 | 18 | 18
mg/L
  Intensive PK (Week 1 or 2) (Cmax): number analyzed (Participants) | 15 | 18 | 15
  Intensive PK (Week 1 or 2) (Cmax) | 0.389 (30.3) | 0.481 (48.9) | 0.369 (57.2)
  Week 8 (Cmax) | 0.180 (37.2) | 0.260 (32.2) | 0.216 (52.6)
  Week 24 (Cmax): number analyzed (Participants) | 17 | 18 | 17
  Week 24 (Cmax) | 0.206 (38.2) | 0.282 (29.0) | 0.248 (44.6)

16. Secondary Outcome: Geometric Mean of Trough Concentration (Ctrough) Bedaquiline
Description: PK parameter determined from plasma concentration-time profiles, dosing information and participant covariates using the final population PK model.
  Lowest concentration at end of the dosing interval which is approximately 24h after dose at Intensive PK (Week 1 or 2) and 48-72h at Weeks 8 and 24.
Time Frame: Intensive PK (Week 1 or 2) 24h post dose and Weeks 8 and 24 48-72h post dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Cohort 1 (≥ 6 to < 18 Years) | Cohort 2 (≥ 2 to < 6 Years) | Cohort 3 (≥ 0 to < 2 Years)
Number analyzed (Participants) | 18 | 18 | 18
mg/L
  Intensive PK (Week 1 or 2): number analyzed (Participants) | 15 | 18 | 15
  Intensive PK (Week 1 or 2) | 0.774 (75.1) | 1.27 (36.7) | 1.07 (79.8)
  Week 8 | 0.356 (61.2) | 0.596 (23.1) | 0.650 (62.5)
  Week 24: number analyzed (Participants) | 17 | 18 | 17
  Week 24 | 0.792 (86.2) | 0.949 (38.3) | 0.935 (60.1)

17. Secondary Outcome: Geometric Mean of Trough Concentration (Ctrough) Bedaquiline Mono-desmethyl Metabolite (M2)
Description: as for outcome 16
Time Frame: Intensive PK (Week 1 or 2) 24h post dose and Weeks 8 and 24 48-72h post dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Cohort 1 (≥ 6 to < 18 Years) | Cohort 2 (≥ 2 to < 6 Years) | Cohort 3 (≥ 0 to < 2 Years)
Number analyzed (Participants) | 18 | 18 | 18
mg/L
  Intensive PK (Week 1 or 2): number analyzed (Participants) | 15 | 18 | 15
  Intensive PK (Week 1 or 2) | 0.381 (31.6) | 0.465 (52.1) | 0.351 (58.6)
  Week 8 | 0.160 (43.6) | 0.236 (33.4) | 0.189 (59.0)
  Week 24: number analyzed (Participants) | 17 | 18 | 17
  Week 24 | 0.196 (40.3) | 0.270 (30.2) | 0.232 (46.8)

18. Secondary Outcome: Median of Time of Maximal Concentration (Tmax) Bedaquiline
Description: as for outcome 15
Time Frame: Intensive PK (Week 1 or 2) pre-dose and 2, 4, 6, 8 hours post dose
Population: as for outcome 7
Measure: Median (Full Range); unit: h
Arm/Group | Cohort 1 (≥ 6 to < 18 Years) | Cohort 2 (≥ 2 to < 6 Years) | Cohort 3 (≥ 0 to < 2 Years)
Number analyzed (Participants) | 15 | 18 | 15
h | 5.91 [3.16 to 6.58] | 5.08 [3.09 to 6.88] | 5.74 [4.03 to 6.98]

19. Secondary Outcome: Median of Time of Maximal Concentration (Tmax) Bedaquiline Mono-desmethyl Metabolite (M2)
Description: as for outcome 15
Time Frame: Intensive PK (Week 1 or 2) pre dose and 2, 4, 6, 8 hours post dose
Population: as for outcome 7
Measure: Median (Full Range); unit: h
Arm/Group | Cohort 1 (≥ 6 to < 18 Years) | Cohort 2 (≥ 2 to < 6 Years) | Cohort 3 (≥ 0 to < 2 Years)
Number analyzed (Participants) | 15 | 18 | 15
h | 0 [0 to 24.3] | 13.4 [0 to 24.2] | 13.6 [0 to 24.3]

20. Secondary Outcome: Geometric Mean of Oral Clearance (CL/F) Bedaquiline
Description: Individual clearance (CL) relative to bioavailability (F) determined from plasma concentration-time profiles, dosing information and participant covariates using the final population PK model
Time Frame: Week 24
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Cohort 1 (≥ 6 to < 18 Years) | Cohort 2 (≥ 2 to < 6 Years) | Cohort 3 (≥ 0 to < 2 Years)
Number analyzed (Participants) | 17 | 18 | 17
L/h | 3.22 (58.0) | 1.45 (35.2) | 1.03 (62.0)

21. Secondary Outcome: Geometric Mean of Theoretical Steady State AUC (AUC0-168h)
Description: Calculated PK parameter determined from weekly continuation phase dose divided by oral clearance at week 24
Time Frame: Week 24
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*mg/L
Arm/Group | Cohort 1 (≥ 6 to < 18 Years) | Cohort 2 (≥ 2 to < 6 Years) | Cohort 3 (≥ 0 to < 2 Years)
Number analyzed (Participants) | 17 | 18 | 17
hour*mg/L | 140 (42.6) | 207 (35.2) | 259 (68.7)

22. Secondary Outcome: Quantitative Post-treatment Bedaquiline Concentrations
Description: as for outcome 15
Time Frame: Weeks 32-96
Reporting Status: Not Posted, anticipated posting 2026-08

23. Secondary Outcome: Post-treatment Bedaquiline Concentrations Below Limit of Quantifications
Description: as for outcome 15
Time Frame: Weeks 32-96
Reporting Status: Not Posted, anticipated posting 2026-08

ADVERSE EVENTS:
Time Frame: From entry through the primary completion date, an average of 76 weeks.
Description: An adverse event (AE) is any unfavorable and unintended sign, symptom, or diagnosis that occurs in a study participant during the conduct of the study REGARDLESS of the attribution. Adverse events are graded on a scale from 1-5: 1=mild, 2=moderate, 3=severe, 4= potentially life-threatening, 5=death. AE grading was per Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table V2.1.
Groups:
- Cohort 1: >= 6 to < 18 Years: Participants ≥30 kg:
  400 mg once per day through the intensive PK sampling visit, then 200 mg three times per week on Monday, Wednesday, and Friday through the Week 24 visit
  Participants ≥15 to <30 kg:
  200 mg once per day through the intensive PK sampling visit, then 100 mg three times per week on Monday, Wednesday, and Friday through the Week 24 visit
- Cohort 2: >= 2 to < 6 Years: Participants >7 to <30 kg:
  200 mg once per day through the intensive PK sampling visit, then 100 mg three times per week on Monday, Wednesday, and Friday through the Week 24 visit
- Cohort 3: >= 0 to < 2 Years: Participants >7 to <30 kg:
  200 mg once per day through the intensive PK sampling visit, then 100 mg three times per week on Monday, Wednesday, and Friday through the Week 24 visit
  Participants ≥ 3 to ≤ 7 kg:
  100 mg once per day through the intensive PK sampling visit, then 50 mg three times per week on Monday, Wednesday, and Friday through the Week 24 visit Hide hide All-Cause Mortality Cohort 1: >= 6 to < 18 Years Cohort 2: >= 2 to < 6 Years Cohort 3: >= 0 to < 2 Years Affected / at Risk (%) Affected / at Risk (%) Affected / at Risk (%) Total 1/18 (5.56%) 0/18 (0%) 0/18 (0%)
Arm/Group | Cohort 1: >= 6 to < 18 Years | Cohort 2: >= 2 to < 6 Years | Cohort 3: >= 0 to < 2 Years
All-Cause Mortality (participants affected / at risk) | 1/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 5/18 | 2/18 | 4/18
Other Adverse Events (participants affected / at risk) | 18/18 | 18/18 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: >= 6 to < 18 Years (N=18) | Cohort 2: >= 2 to < 6 Years (N=18) | Cohort 3: >= 0 to < 2 Years (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis viral (Infections and infestations) | 0 | 0 | 1
Infective exacerbation of asthma (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Otitis media staphylococcal (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0
Childhood asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: >= 6 to < 18 Years (N=18) | Cohort 2: >= 2 to < 6 Years (N=18) | Cohort 3: >= 0 to < 2 Years (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 2 | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 2 | 0
Conductive deafness (Ear and labyrinth disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 0 | 0
Teething (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 8 | 4 | 2
Chest pain (General disorders) | 2 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 3 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0
Immune reconstitution inflammatory syndrome (Immune system disorders) | 1 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 2
Hepatitis A (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 2 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 3
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0
Pustule (Infections and infestations) | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Tinea capitis (Infections and infestations) | 1 | 2 | 2
Tinea versicolour (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 0
Urethritis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Viral tonsillitis (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 7 | 7 | 4
Aspartate aminotransferase increased (Investigations) | 8 | 11 | 7
Bilirubin conjugated increased (Investigations) | 2 | 0 | 1
Blood albumin decreased (Investigations) | 5 | 2 | 4
Blood bicarbonate (Investigations) | 0 | 0 | 1
Blood bicarbonate decreased (Investigations) | 18 | 18 | 17
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood calcium decreased (Investigations) | 2 | 1 | 3
Blood calcium increased (Investigations) | 1 | 3 | 9
Blood creatinine increased (Investigations) | 9 | 12 | 11
Blood lactic acid abnormal (Investigations) | 11 | 0 | 1
Blood magnesium decreased (Investigations) | 8 | 1 | 2
Blood phosphorus decreased (Investigations) | 0 | 0 | 1
Blood potassium decreased (Investigations) | 2 | 1 | 0
Blood potassium increased (Investigations) | 9 | 5 | 12
Blood pressure diastolic increased (Investigations) | 0 | 0 | 5
Blood pressure increased (Investigations) | 0 | 1 | 2
Blood pressure systolic increased (Investigations) | 0 | 2 | 1
Blood sodium decreased (Investigations) | 7 | 14 | 15
Blood sodium increased (Investigations) | 2 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0
Carbon dioxide decreased (Investigations) | 1 | 0 | 2
Haemoglobin decreased (Investigations) | 9 | 13 | 9
Neutrophil count decreased (Investigations) | 6 | 5 | 8
Platelet count decreased (Investigations) | 2 | 1 | 3
Weight decreased (Investigations) | 2 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 0
Underweight (Metabolism and nutrition disorders) | 7 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Blount's disease (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Vulvovaginal warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 6
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pityriasis alba (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 | 3 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Systolic hypertension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights

DOCUMENTS (4):
  • Study Protocol and Informed Consent Form: Protocol and ICF (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT02906007/Prot_ICF_000.pdf
  • Study Protocol: Letter of Amendment #1 (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/07/NCT02906007/Prot_001.pdf
  • Study Protocol: Clarification Memorandum #1 (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/07/NCT02906007/Prot_002.pdf
  • Statistical Analysis Plan (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT02906007/SAP_003.pdf